CLINICAL TRIAL: NCT02703168
Title: Post-marketing Study to Document Long-term Performance of Straumann Tissue Level Implants With SLActive Surface in the Posterior Mandible and Maxilla After Immediate or Early Loading - Follow-up to Study CR 06/03
Brief Title: Long-term Performance of SLActive Implants After Immediate or Early Loading
Status: Completed | Type: Observational
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Other Study IDs: CR 03-05/11
Record Dates: First submitted 2015-09-11; First posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Partial Edentulism
Keywords: Dental implants

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Immediate loading: Patients were allocated to treatment group in the core study. Immediate loading was defined as follows: Implant(s) will be restored with a temporary restoration on the day of surgery
- Early loading: Patients were allocated to treatment group in the core study. Early loading was defined as follows: Healing caps will be placed on the implant(s) immediately after surgery. A provisional restoration will be placed between day 28 to day 34 post surgery

SUMMARY:
This is a follow-up study with patients, who participated in the Straumann clinical study CR06/03. The objective is the assessment of long-term data (8 and 10 years after implantation) on the performance of immediate and early (28-34 days post implantation) non-occlusal loaded Straumann Tissue Level Implants with SLActive surface when used to support single crowns or 2-4 unit fixed dental prostheses in the posterior maxilla and mandible.

The primary objective is of the study is to analyse the change in crestal bone levels 8 and 10 years post-surgery compared to 6 months, 1 year, 2 years and 3 years post-surgery in the immediate and early loading group.

DETAILED DESCRIPTION:
This is a prospective, post-market, open label, follow-up multicenter study with patients who participated in the Straumann clinical study CR06/03. The total study duration for each patient should be 2 years.

In total 2 visits are scheduled in this study. Bone level changes, implant success and survival, performance of the restorative components, and adverse events (AEs) will be assessed.

The study device is a CE-marked product and FDA approved.

Three centres, one in Portugal and two in Germany, will participate.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent
* Patients with Straumann SLActive tissue level implants, who participated in the Straumann CR06/03 clinical study.
* Patients must be committed to the study for its full duration.
* Patient's Radiographic stent must be available from study CR06/03

Exclusion Criteria:

* Use of any investigational drug or device within 30 days before start of the study.
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with the analysis of the study results, such as history of non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who participated in the Straumann clinical trial CR06/03
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2012-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Crestal bone level change by radiographic assessment | 8 and 10 year post-surgery
  To evaluate the changes in crestal bone levels (in millimetre) in relation to defined implant reference point and different time points (between baseline at implant insertion and follow-up time points at 8 and 10 years after implant insertion) in the maxilla and mandible of the immediate and early loading groups.

SECONDARY OUTCOMES:
Implant survival by clinical and radiographic assessment | 8 and 10 year post-surgery
  To evaluate the implant survival rate by clinically and radiographically count of implants still in place in the subject's jaw bone at the time of assessment (8 and 10 years post-surgery). The implant survival rates will be compared between the treatment groups (immediate loading and early loading).
Incidence of adverse events and adverse device effects | 8 and 10 year post-surgery
  Total number of AEs and total number of AEs related to the study treatment (device-related or procedure-related), as well as the total number of subjects affected by at least one adverse event wil be calculated per treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Jackowski, Prof., Principal Investigator — Universität Witten/Herdecke; Tim Krafft, Dr. Dr., Principal Investigator — Kieferchirurgische Praxisgemeinschaft, Weiden; Pedro Nicolau, Dr., Principal Investigator — University of Coimbra

IPD SHARING:
Plan to Share IPD: No